CLINICAL TRIAL: NCT06634563
Title: Effect Of Adding Mindfulness Meditation To Cognitive Behavioral Training On Pain And Quality Of Life In Fibromyalgia
Acronym: CB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Abd el Aziz Abd el Salam, principale investigator dina abd el-aziz, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005340
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Fibromyalgia
Keywords: Mindfulness Meditation; cognitive behavioral training; fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Mindfulness Meditation and cognitive behavioral training
Who Masked: Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mindfulness meditation (Experimental): Twenty five women in study group will receive mindfulness meditation for 30 minutes in addition to mobile application-based brain training program (cognitive behavioral training) for 30 minutes day after day for 8 weeks
  Interventions: Other: mindfulness meditation; Other: cognitive behavioral training
- cognitive behavioral training (Active Comparator): Twenty five women in control group will receives mobile application-based brain training program (cognitive behavioral training) for 60 minutes day after day for 8 weeks.
  Interventions: Other: cognitive behavioral training

INTERVENTIONS:
Other: mindfulness meditation — the patients will receive mindfulness meditation in the form of Attention-focusing technique (body scan, directing attention throughout the body in a relaxed, supine state) guided by audiotapes. Relaxing every part of the body by guided audiotape from head to toes and Sitting meditation (systematically directing attention to breath) guided by audiotapes. Relaxing deep rhythmic breathing with concentration on every breath.
  Arms: mindfulness meditation
Other: cognitive behavioral training — Training sessions will include three cognitive training tasks each of them target a particular core cognitive capability and are grouped into three categories by target domain: memory (working memory), attention (selective attention), and problem solving (logical reasoning) through these games (organic order and fuse clues for logical reasoning training, lost in migration, trouble brewing, assist ants and train of thought for attention training and memory match and memory match one drive for working memory training).

SUMMARY:
this study will be conducted to investigate The Impact Of Adding Mindfulness Meditation to Cognitive Behavioral Training On Pain And Quality Of Life In Fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FMS) is a disorder characterized by chronic, widespread musculoskeletal pain. Muscle and joint stiffness, insomnia, fatigue, mood disorders, cognitive dysfunction, anxiety, and generalized sensitivity are the main manifestations of this disease .Cognitive-behavioral training presents as an important therapeutic resource, as it is capable of modifying patient's negative thoughts and expectations, improving mood, stress, coping with pain and problem solving, including behavioral interventions that specifically deal with improving the fibromyalgia symptoms (sleep hygiene, re-laxation training, activity rhythm).Mindfulness meditation is the intentional effort to pay nonjudgmental attention to present-moment experiences and sustain this attention over time. The aim is to cultivate a stable and nonreactive present-moment awareness. Mindfulness Based Pain Management has been evaluated and showing significant positive changes in patients with chronic pain, with medium to large effect sizes on self-report measures of depression, positive outlook, pain acceptance. fifty women with fibromylagia will be assigned randomly to two groups; first one will receive mindfulness meditation for 30 minutes in addition to mobile application-based brain training program and the second one will receive mobile application-based brain training program alone

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of a clinical diagnosis of fibromyalgia by the patient's own physician.
* Wide spread pain for at least 3 months and tenderness at a minimum of 11of the 18 specific tender point sites.
* Age between 30 and 40 years.
* Female gender.
* BMI: 25-30 kg/m2

Exclusion Criteria:

* Pregnancy
* drug addicition
* Any current psychiatric disorder that would interfere with pro-gram adherence.
* Life-threatening disease

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-12 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
pressure threshold | up to eight weeks
  The algometer with a rubber disc of 1 cm2 will be applied at a 90° vertical angle to all 18 tender point. Previous studies have shown pressure threshold measures obtained using algometer with 1 cm2 contact area to have acceptable interrater and intrarater reliability of pressure scores over time. Pressure will be steadily increased at a rate of approximately 1 kg per second, and each site will be tested in succession for each of two trials, allowing for recovery time between trials (approximately 10 minutes between retest at each point). Subjects will be instructed to indicate verbally when they first felt pain. The pressure will be then stopped, and the pressure will be recorded
severity of pain | up to eight weeks
  The Visual Analogue Scale-Pain (VAS-Pain) will be used to assess pain. the patients will be asked to assess the severity of pain they experience at that moment on a 10-cm visual scale from 0 (no pain) to 10 (the most painful possible).
cognition assessment | up to eight weeks
  Reha-Com device will be used to assess cognition. it containing the (attention and concentration) program was utilized as the patient is asked to concentrate on every detail in the separately presented picture and select the one that resembles it in every detail from the matrix, as the assessment screen is splitted into two parts. One portion represents the matrix that involves: according to (24) levels of difficulty: 3 pictures (1 by 3 matrix), 6 pictures (2 by 3 matrix) as well as 9 pictures (3 by 3 matrix), and the other part represents the separated picture. Reha-Com devicealso containing the (Memory) program. The test is divided into three different "modules" according to levels of difficulty. Every module is represented by a distinct task the "player" is asked to perform: memorizing all cards (Storage systems), memorizing cards selectively (Selective attention) and sorting cards (Central executive).

SECONDARY OUTCOMES:
life disability | up to eight weeks
  The revised Fibromyalgia Impact Questionnaire will be used to assess quality of life. It consists of 21-items, 11-point numerical rating scales (0-10) designed to evaluate three main domains in relation to the previous week: physical function (9 items), overall impact (2 items) and FM symptoms (10 items). It is also available in arabic version. The Arabic version of the FIQ-A has an acceptable reliability and validity criteria. It can be used for clinical practice and research use in the Arabic-speaking population